CLINICAL TRIAL: NCT06447064
Title: Cancer Loyalty Card Study 2: a Retrospective Observational Case-Control Study
Brief Title: Cancer Loyalty Card Study 2 (CLOCS-2)
Acronym: (CLOCS-2)
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: University of Birmingham (Other); University of Nottingham (Other); University of Central Lancashire (Other); Cancer Research UK (Other); Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 324742
Record Dates: First submitted 2024-06-03; First posted 2024-06-06 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer; Colon Cancer; Oesophageal Cancer; Stomach Cancer; Liver Cancer; Bladder Cancer; Uterine Cancer; Vulvar Cancer; Ovarian Cancer; Endometrial Cancer
Keywords: Ovarian Cancer; Epidemiology; Observational Study; Risk Assessment
MeSH Terms: conditions — Pancreatic Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Liver Neoplasms; Urinary Bladder Neoplasms; Uterine Neoplasms; Vulvar Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Participants diagnosed with cancer.
  Interventions: Other: Cases & Controls
- Controls: Participants not diagnosed with cancer.
  Interventions: Other: Cases & Controls

INTERVENTIONS:
Other: Cases & Controls — Participants will complete a brief online questionnaire at REDCap about their health, clinical history and lifestyle choices. The participant will only need to provide a photo ID and utility bill for ID verification, if the retailer cannot match participant details. After recruitment the participants purchase history in the past 6 years will be requested from the retailers.

SUMMARY:
Cancer is one of the leading causes of mortality worldwide and is responsible for an estimated 9.6 million deaths yearly. Cancer-related deaths can be reduced if patients are diagnosed and treated early. Delay in cancer diagnosis can occur at any point along the diagnostic spectrum, from the first observation of symptoms to the start of treatment. Diagnosing cancer when it is still at an early stage, before it has spread, gives surgery, radiotherapy and other treatments the best chance of working.

Therefore, early diagnosis is the most important way to improve cancer outcomes.Most of the cancers usually presents with vague and non-alarming symptoms. Most individuals are diagnosed late when the cancer has already spread, and the prognosis is poor. There are over 200 different types of cancer that can cause many different signs and symptoms. Sometimes symptoms affect specific body areas, such as abdomen or skin. But signs can also be more general, and include weight loss, tiredness (fatigue) or unexplained pain. The type of symptoms varies from person to person.

The major reasons for not presenting to the GP with symptoms such as these are "not wanting to waste the GP's time" and normalisation of these symptoms.

The persistence of a symptom, social influence and awareness encourage help-seeking behaviours in primary care. However, few believe their symptom(s) might be a sign of cancer. Consequently, people might choose to self-manage their symptoms by using over-the-counter medication, and to seek advice from other sources, (pharmacists, family, internet), rather than a primary care physician.

RATIONALE FOR CURRENT STUDY

An early cancer diagnosis is essential for receiving treatment as early as possible to have the best chance for successful treatment. Early diagnosis of cancer can be challenging. Sometimes, the cancer symptoms resemble common illnesses and could resolve with the use of over-the-counter medications and other remedies until they become persistent or debilitating. The present study focuses on ten cancer forms: colon, oesophageal, stomach, liver, bladder, uterine, vulval, ovarian, endometrial and pancreatic. Patients diagnosed with the cancers mentioned above often report experiencing vague symptoms (such as abdominal or back pain, indigestion, feeling full etc). They often use over-the-counter medication to manage their symptoms before seeing a doctor.

Information about how often and what products participants purchase (e.g. pain killers, digestive products and natural remedies) to care for these symptoms could help identify these cancers a few crucial weeks or months earlier and encourage people to seek help sooner from their doctors.

DETAILED DESCRIPTION:
Purpose and Design

The Cancer Loyalty Card Study-2 (CLOCS-2) addresses whether or not data already collected by high street retailers can detect significant changes in cancer patients' purchase behaviours before their diagnosis. The aim is to conduct a case-control study of cancer patients matched with participants without these cancer types. 1450 recently diagnosed cancer patients and 1450 participants as controls will be recruited and up to six years of prior purchase data will be collated.

Recruitment

Participants, 18 years or older, with any of the aforementioned cancer forms and having at least one of the participating high street retailer's loyalty cards from Tesco or Boots in their household, will be recruited through the GP invites, NHS cancer clinics and Be Part of Research.

All participants registering in the study and not holding the primary ownership of the loyalty cards from Tesco or Boots must register in the study along with the primary owner of the loyalty card from the same household. All the collected data will be safeguarded in a secure enclave with limited access to the CLOCS-2 team.

Consent

All participants will be given the information sheet and consent form through a REDCap link shared through messages sent by GP, cancer clinics or Be Part of Research. They can take as much time as they need to read through the information sheet. If they choose to participate, they can complete the consent form whenever convenient and fill it out online at REDCap.

Methods

Loyalty card holders with primary ownership of at least one of the participating high street retailers loyalty cards from Tesco or Boots and their family members living in the same household are eligible to participate in CLOCS-2. All participants will be invited to join the study by invites (sent through text messages from GP, cancer clinics or Be Part of Research) and can choose to sign up via a link provided in invites that leads to REDCap. People over 18 years of age and with any form of cancer as listed earlier and who use at least one of the participating high street retailer's loyalty cards in their household will be recruited as cases. Whereas people over 18 years of age, without the diagnosis of these cancer types and using at least one of the participating high street retailer's loyalty cards in their households will be recruited as control participants.

Consenting participants will complete a brief online questionnaire at REDCap about their health, clinical history and lifestyle choices. To adhere to participating high street retailers' policies, only participants whose details cannot be matched to that of the retailers' will need to provide a photo ID and utility bill for ID verification.

The tentative participant recruitment date is 01/11/2025. Once the participants are recruited in the study, their past six years of purchase history will be requested from Tesco/Boots from the recruitment date. This data received from these high street retailers will be non-identifiable pseudonymised data. Participant identity will be linked to the analysis datasets only through a unique barcode assigned when completing the recruitment questionnaire, meaning the data will be pseudonymised. The only identifiable information will be on the consent form and the participant barcode. Retailer and questionnaire data will only be linked via the pseudonymised participant barcode.

If participants consent to be re-contacted by the CLOCS-2 team for future studies or loyalty card detail clarification, they can opt for it in their consent forms. No further action is needed from participants once they complete their consent form and questionnaire (and clarify loyalty card details if necessary). Participants will be provided with the study's website and encouraged to visit the study's website for updates.

ELIGIBILITY:
Inclusion Criteria (ALL):

* Individuals aged >18 years of age
* Individuals must be residing in the United Kingdom at the time of giving informed consent
* Individuals must be registered with an NHS GP Practice
* Individuals must meet the criteria of ONE of the groups. For example, to be eligible for Group 1 (Cases), individuals must have been diagnosed with one of the following cancer types in the last 24 months: Bladder, colorectal (bowel), endometrial, liver, oesophageal, ovarian, pancreatic, stomach (gastric), uterine, or vulval; whereas for Group 2 (Controls), individuals must not have received a cancer diagnosis of any type in the last 6 years (except where the diagnosis was of non-melanoma skin cancer).
* Individuals must be a primary registered cardholder* of one of the loyalty cards listed below, and consent to share their loyalty card data with the study team
* Tesco Clubcard
* Boots Advantage Card
* Provision of written informed consent
* Willing and able to comply with all required study activities

  * The primary registered card holder, i.e., the person who is named on the loyalty card account, must also enrol into the study, if someone other than the registered primary card holder from the same household, wants to take part in the study.

Exclusion Criteria (ALL):

* Individuals under the age of 18 years
* Non-UK residents, at the time of giving informed consent
* Individuals without an eligible loyalty card, or who have no one in their household who has an eligible loyalty card
* Individuals who are not the primary registered cardholder in their household and where the primary registered loyalty card holder is not willing to join the study, and/or where the primary registered cardholder does not make purchases for or on behalf of the individual

Exclusion Criteria (CASES):

• Individuals will not be able to join as a case if:

* they have been diagnosed with an eligible cancer type more than 24 months ago (except where the diagnosis was non-melanoma skin cancer).
* they have received an ineligible cancer diagnosis within the last 6 years except where the diagnosis was non-melanoma skin cancer).

Exclusion Criteria (Controls):

• Individuals will not be able to join as a control (Group 2) if:

o they have received any cancer diagnosis in the last six years (except where the diagnosis was non-melanoma skin cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged ≥18 years old, who own at least one participating high street retailer loyalty cad in their household. Among these individuals, those who have been diagnosed with any form of cancer as mentioned above (can join the CLOCS-2 as cases, and those who have no prior cancer diagnosis from the list of cancers mentioned above are eligible to join as controls.
Sampling Method: Probability Sample
Enrollment: 2900 (Estimated)
Dates: Start 2026-01-29 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Purchase behaviours (purchase of pain relief medications) assessed by Statistical Model | 3 years
  The primary outcome of the CLOCS-2 will be to define the time by which the cases and controls are statistically significantly (p≤0.05) different in their purchase behaviours leading up to a cancer diagnosis on a population level.

SECONDARY OUTCOMES:
Alert about Cancer symptoms assessed by purchase behaviour | 3 years
  Defining a purchase threshold as an 'alert' about cancer symptoms in individuals and determining the predictive utility of purchasing behaviours in the early detection of these cancer forms.
Development of risk profiles for each cancer type | 3 years
  Risk profiles for each main cancer type created from the participants self-reported health data; adjusted for in the analyses
Development of predictive model to assess utility of purchasing behaviours | 3 years
  A predictive model to assess the utility of identified purchasing behaviours in early cancer detection, tested for efficacy of its predictive utility of purchasing behaviours in the early detection of these cancer forms

CONTACTS AND LOCATIONS:
Overall Officials: Dr James Flanagan, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only aggregated and anonymised survey data will be shared with other researchers after publication. No sensitive individual level data will be shared.